CLINICAL TRIAL: NCT05426551
Title: Validation of the Dual-isotope Method for Measuring Ileal Protein Digestibility
Acronym: VALDIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: St. John's Research Institute (Other)
Responsible Party: Principal Investigator, Robert Benamouzig, Professor, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VALDIM
Record Dates: First submitted 2022-05-31; First posted 2022-06-22 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: amino acid digestibility; dual isotope method; labelled protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bolus-spi (Experimental): The volunteers will consume the test-meal as a bolus in one time at t = 0, with 13C-spirulina as the reference protein
  Interventions: Other: Dual isotope method
- Plateau-spi (Experimental): The volunteers will consume the test-meal in a plateau feeding protocol, with 13C-spirulina as the reference protein
  Interventions: Other: Dual isotope method
- Plateau-AA (Experimental): The volunteers will consume the test-meal in a plateau feeding protocol, with 13C-free AA mixture as the reference "protein"
  Interventions: Other: Dual isotope method

INTERVENTIONS:
Other: Dual isotope method — The digestibility of amino acids will be determined within each arm by the collection of ileal digesta owing to naso-ileal intubation device and by plasma samples with the dual isotope method.

SUMMARY:
The dual isotope method has been recently developed and used to evaluate indispensable amino acid (IAA) digestibility of various protein food such as legumes, eggs and chicken meat in healthy adults and children. The dual isotope method is an indirect method based on the measurement in plasma of absorbed IAA from a deuterium (2H) intrinsically labeled test protein compared against the same IAA of a carbon 13 (13C) intrinsically labeled standard protein of known digestibility or crystalline amino acids (AA) of theoretical 100% digestibility. However, digestibility data estimated with the dual isotope method have not been directly compared with ileal IAA digestibility directly determined through ileal digesta sampling. The goal of this study is to assess the IAA digestibility of intrinsically 2H-hen's egg in healthy volunteers using both indirect and direct methods.

DETAILED DESCRIPTION:
The test meal will consist of 60 g of lyophilized whole egg powder which contains 30 g of 2H-egg protein and 800 mg [U-13C]-spirulina or 400 mg of 13C free AA mixture, mixed with water and cooked as an omelet. The 2H-egg powder has been produced by our collaborators of the St John's Research Institute in Bangalore (India). Celite (acid insoluble ash, Advanced Minerals Corporation) will be added to the meal as an indigestible marker to check the recovery of the meal in effluents. The test-meal will be given as a bolus or in a plateau feeding (repeated mini-meals) depending of the groups of subjects. 600 g of 2H-labeled lyophilized eggs will be obtained from layer hens administered a uniformly 2H-labeled AA mix orally for 60 d with their daily feed. Microbiological analyses will be performed to ensure their safety for human consumption.

18 volunteers will be included at the end of the study and tested at the Human Nutrition Research Centre of Avicenne Hospital (France). The main inclusion criteria are men and women, 18 to 45 year-old, body mass index (BMI) 18 to 30 kg/m2. The main exclusion criteria are any digestive or hepatic pathology, allergy against eggs, allergy against latex, pregnant women. Due to the invasive procedure of intubation, the investigators plan to recruit 30 volunteers to accommodate for the usual 40% dropouts.

The subjects will be divided in 3 groups of n = 6:

* Bolus-spi, n = 6, the volunteers will consume the test-meal as a bolus in one time at t = 0, with 13C-spirulina as the reference protein
* Plateau-spi, n = 6, the volunteers will consume the test-meal in a plateau feeding protocol, with 13C-spirulina as the reference protein
* Plateau-AA, n = 6, the volunteers will consume the test-meal in a plateau feeding protocol, with 13C-free AA mixture as the reference "protein"

One week before the experiment, the volunteers will follow a standard diet adapted to their body weight to control their protein intake (1.3 g protein/kg body weight).

The volunteers will arrive at the Human Nutrition Research Centre of Avicenne Hospital on the morning before the day of the experiment. They will be equipped with a triple lumen intestinal tube that will be allowed to progress through the intestinal tract for 24 h. One of the lumen is radio opaque and serves to perfuse a non-absorbable maker in the intestine (slow marker method). The second lumen is dedicated to inflate a weighted balloon that facilitate the migration of the tube. The third lumen is dedicated to the continuous aspiration of the effluents, 15 cm below the perfusion site. The measurement of the non-absorbable marker in the effluents allows the determination of the effluent flow rate.

On the day of the experiment, the position of the tube will be checked by radiography to verify its location at the terminal ileum. A catheter will be inserted in the forearm vein for blood sampling. The perfusion of the non-absorbable marker, polyethylene glycol (PEG) 4000 (20 g/l), will start at a flow rate of 1 ml/min. The intestinal flow and the basal ileal sample will be collected during 30 min. Basal plasma and urine sample will be collected.

At t = 0, the volunteers of the group "Bolus-spi" will consume all the test-meal in less the 20 min. For the volunteers of the groups "Plateau-spi" and "Plateau-AA", the test-meal will be divided into 22 equal portions and they will consume the first meal as a priming dose of 6 mini-portions. Then, they will consume single mini-portions every 30 min for 7.5 h. One portion will be dedicated to meal analyses. Until t = 8, intestinal content will be continuously collected by aspiration and pooled every 30 min. Blood will be sampled hourly during 4 h and every 30 min from t = 5 to t = 8. Urine will be collected every 2 h until t=8 (total volume of urine output will be noted at each time point for proportional pooling). Breath samples will be collected every 30 min. Carbon dioxide output (VCO2) will be evaluated hourly during 10 min by indirect calorimetry (Canopy). Urine sample will be collected at the start of the experiment and during the study protocol. Fecal samples will be collected before the start of the experiment and within the next 24 h. The naso-ileal tube will be removed after the last collection of effluent at t = 8.The naso-ileal tube will be removed after the last collection of effluent at t=8.

The following analyses will be performed:

* Concentration of PEG-4000 by turbidimetric method in digesta samples
* Total hydrogen content and 2H enrichment in meals and digesta samples by isotope-ratio mass spectrometry (IRMS) coupled to pyrolysis analyzer
* Total carbon content and 13C enrichment in meals and digesta samples by Elemental analyzer (EA) coupled to IRMS
* AA concentration in meals and digesta samples by Ultra High Performance Liquid Chromatography (UHPLC)
* 13C-AA and 2H-AA enrichment plasma and meal samples by Liquid Chromatography coupled to tandem Mass Spectrometry (LC-MS/MS)
* 13C-AA and 2H-AA enrichment in digesta and meal samples by gas chromatography-combustion-isotope ratio mass spectrometry (GC-C-IRMS)
* Celite content in pooled (0-8 h) digesta samples
* 13CO2 in breath sample by Multiflow-IRMS
* Amino-acidome and peptidome of digesta, plasma, urine, and fecal samples

Part of the analyses (13C-AA and 2H-AA enrichment plasma and meal by LC-MS/MS, -omic analyses) will be done by our collaborators of the St John's Research Institute in Bangalore (India).

ELIGIBILITY:
Inclusion Criteria:

* 18<BMI<30
* Healthy
* Insured under the French social security system
* For women: use of birth control
* Signed informed consent

Exclusion Criteria:

* Any dietary allergy
* Latex allergy
* Positive serology to HIV, hepatite C virus antibody, hepatite B virus surface antigen and core antibodies
* Gluten intolerance
* Anemia
* Use of drugs
* High consumption of alcohol
* Hypertension, diabetes, digestive disease, hepatic or renal disease, severe cardiac disease
* Pregnancy
* High sport practicing (>7h/wk)
* Blood donation in the 3 months prior to the study
* Participation in a clinical study in the 3 months prior to the study
* No signed informed consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-10-23 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Real ileal amino acid digestibility | -30 minute to 8 hours after the first meal
  The measurements of amino acid concentration (mmol) and their individual 2H enrichment (atom %) allow the determination of dietary amino acids remaining in the lumen.
  Dietary amino acids that are recovered in the ileal samples are then considered as non absorbed and expressed as % of amino acid ingested, it allows the calculation of real ileal amino acid digestibility (100 - dietary amino acid not absorbed)
Indirect amino acid digestibility | -30 minute to 8 hours after the first meal
  The individual amino acid 2H enrichment (atom %) and 13C enrichment (atom %) in the meal and in the plasma from 5 h to 8 h or 0 h to 8 h after the first meal (depending of the group) will be evaluated to calculate their ratio:
  Ratio meal AAi = 2H meal AAi / 13C meal AAi Ratio plasma AAi = 2H plasma AAi / 13C plasma AAi
  The ratio of the meal and plasma ratios will be corrected by the known digestibility of spirulina amino acid or free amino acid (in %, depending of the group) to determine the indirect amino acid digestibility of lyophilized egg protein with the following formula:
  Indirect ileal amino acid digestibility (%) = AAi ileal digestibility spirulina or free AA mix (%) x Ratio plasma AAi / Ratio meal AAi

SECONDARY OUTCOMES:
Urinary, fecal and plasma individual amino acid concentration in response to protein ingestion | -30 minute to 8 hours after the first meal
  Determination of amino acids concentrations (in mmol) in plasma, urinary and fecal samples and bioinformatic analysis, before and after ingestion of protein meal for characterisation of non- or minimally-invasive markers of digestibility
Plasma, urinary and fecal peptidome in response to protein ingestion | -30 minute to 8 hours after the first meal
  Sequencing of peptides in plasma, urinary and fecal samples and bioinformatic analysis, before and after ingestion of protein meal for characterisation of non- or minimally-invasive markers of digestibility
Gut microbiota in response to protein ingestion | Before and 24 hours after meal intake
  Microbial DNA sequencing of fecal samples before and after ingestion of protein meal

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche sur Volontaires (CRV) de l'hôpital Avicenne, Bobigny, France